CLINICAL TRIAL: NCT04876391
Title: An Open-label, Long-term Extension Trial of Spesolimab Treatment in Adult Patients With Hidradenitis Suppurativa (HS)
Brief Title: A Study Investigating Long-term Treatment With Spesolimab in People With a Skin Disease Called Hidradenitis Suppurativa Who Completed a Previous Clinical Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1368-0067; 2020-005587-55 (EudraCT Number)
Record Dates: First submitted 2021-05-04; First posted 2021-05-06 (Actual); Results first posted 2025-06-08 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Hidradenitis Suppurativa
MeSH Terms: conditions — Hidradenitis Suppurativa | interventions — spesolimab

STUDY DESIGN:
Masking Description: All medication kit assignments will occur in an open label fashion except for medications provided for visit 1. Only administration of study medication at visit 1 is blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Prior Placebo (PP) (Experimental): Participants in the placebo arm of the 1368-0052 Proof of Concept Clinical (PoCC) trial received an initial 1200 mg intravenous (i.v.) loading dose of spesolimab plus subcutaneous (s.c.) placebo at Visit 1, followed by 600 mg s.c. doses of spesolimab every two weeks for the next 12 weeks. Further dosing was based on changes in HS-PGA grade assessment from baseline to week 12.
  Interventions: Drug: Spesolimab 1200 mg; Drug: Spesolimab 600 mg; Drug: Placebo matching 600 mg Spesolimab
- Prior Spesolimab (PS) (Experimental): Participants in the active arm of the 1368-0052 Proof of Concept Clinical (PoCC) trial received an initial 600 mg subcutaneous (s.c.) loading dose of spesolimab plus intravenous (i.v.) placebo at Visit 1, followed by 600 mg s.c. doses of spesolimab every two weeks for the next 12 weeks. Further dosing was based on changes in HS-PGA grade assessment from baseline to week 12.
  Interventions: Drug: Spesolimab 600 mg; Drug: Placebo matching 1200 mg Spesolimab

INTERVENTIONS:
Drug: Spesolimab 1200 mg — Participants in the 1368-0052 PoCC trial's placebo arm received a 1200 mg intravenous (i.v.) loading dose at Visit 1, then 600 mg s.c. every two weeks for 12 weeks.
  Arms: Prior Placebo (PP)
Drug: Spesolimab 600 mg — Participants in the 1368-0052 PoCC trial's active arm received a 600 mg subcutaneous (s.c.) loading dose of spesolimab at Visit 1, followed by 600 mg s.c. every two weeks for 12 weeks.
Drug: Placebo matching 600 mg Spesolimab — Participants from the placebo arm of the 1368-0052 PoCC trial will receive a subcutaneous (s.c.) administration of placebo matching 600 mg spesolimab at Visit 1.
  Arms: Prior Placebo (PP)
Drug: Placebo matching 1200 mg Spesolimab — Participants from the active arm of the 1368-0052 PoCC trial will receive an intravenous (i.v.) infusion of placebo matching 1200 mg spesolimab at Visit 1
  Arms: Prior Spesolimab (PS)

SUMMARY:
This study is open to adults with hidradenitis suppurativa who took part in a previous clinical study of a medicine called spesolimab. Participants who completed treatment can join this study.

The purpose of this study is to find out how safe spesolimab is and whether it helps people with hidradenitis suppurativa in the long-term. Participants are in this study for about 2 years and 4 months. For 2 years, participants visit the study site every 2 weeks to get spesolimab injections under the skin. At study visits, doctors check the severity of participants' hidradenitis suppurativa and collect information on any health problems of the participants.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have completed treatment in the parent Hidradenitis suppurativa (HS) spesolimab trial (1368-0052) without premature discontinuation
* Signed and dated written informed consent in accordance with ICH Harmonized Guideline for Good Clinical Practice (ICH-GCP) and local legislation prior to admission to the trial
* Woman of childbearing potential (WOCBP) must be ready and able to use highly effective methods of birth control per ICH M3 (R2) that result in a low failure rate of less than 1% per year when used consistently and correctly. A list of contraception methods meeting these criteria is provided in the patient information and consent form.

Exclusion Criteria:

* Women who are pregnant, nursing, or who plan to become pregnant while in the trial
* Patients who experienced study treatment-limiting adverse events during the 1368-0052 parent trial
* Severe, progressive, or uncontrolled condition such as renal, hepatic, haematological, endocrine, pulmonary, cardiac, neurologic, cerebral, or psychiatric disease, or signs and symptoms thereof
* Any new documented active or suspected malignancy except appropriately treated basal cell carcinoma, squamous cell carcinoma of the skin or in situ carcinoma of uterine cervix
* Use of any restricted medication or any drug considered by the investigator likely to interfere with the safe conduct of the study since the last visit of the 1368-0052 parent trial
* History of allergy/hypersensitivity to the systemically administered trial medication agent or its excipients
* Major surgery (major according to the investigator's assessment) planned during this extension trial (e.g. hip replacement, aneurysm removal, stomach ligation), as assessed by the investigator
* Any condition which in the opinion of the investigator affects the safety of the patient, the patient's ability to participate in this trial or could compromise the quality of data Further exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2021-08-24 (Actual); Primary Completion 2024-04-26 (Actual); Study Completion 2024-04-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (26):
- United States (4):
  - Dermatology Research Associates, Los Angeles, California
  - Dawes Fretzin Clinical Research Group, LLC-Indianapolis-58713, Indianapolis, Indiana
  - Mayo Clinic, Rochester, Rochester, Minnesota
  - Unity Clinical Research, Oklahoma City, Oklahoma
- Australia (2):
  - Holdsworth House Medical Practice, Sydney, New South Wales
  - Royal Melbourne Hospital, Parkville, Victoria
- Cliniques Universitaires Saint-Luc, Brussels, Belgium
- Dr. S. K. Siddha Medicine Professional Corporation, Newmarket, Ontario, Canada
- University Hospital Ostrava, Ostrava, Czechia
- France (3):
  - CLI Reims Bezannes, Bezannes
  - HOP Edouard Herriot, Lyon
  - HOP Larrey, Toulouse
- Germany (3):
  - Katholisches Klinikum Bochum gGmbH, Bochum
  - Städtisches Klinikum Dessau, Dessau
  - Universitätsklinikum Frankfurt, Frankfurt am Main
- Italy (2):
  - Ospedali Riuniti di Ancona, Ancona
  - Azienda Ospedaliera Universitaria Pisana, Pisa
- Erasmus Medisch Centrum-ROTTERDAM-50697, Rotterdam, Netherlands
- Norway (3):
  - Haukeland Universitetssykehus, Bergen
  - Nordlandssykehuset HF, Bodø, Bodø
  - Oslo Universitetssykehus HF, Rikshospitalet, Oslo
- Poland (2):
  - Non-Public Health Care Facility LABDERM, Ossy
  - Cityclinic Medical and Psychological Clinic Matusiak Partnership, Wroclaw
- Spain (3):
  - Hospital Santa Creu i Sant Pau, Barcelona
  - Hospital La Princesa, Madrid
  - Hospital Universitario 12 de Octubre, Madrid

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a multi-national, multi-centre, non-controlled, single-arm, open-label extension trial of the proof-of-clinical-concept (PoCC) trial 1368-0052, consisting of a 104-week treatment period and a 16-week safety follow-up. Patients from the PoCC trial (spesolimab or placebo group) rolled over into this trial. The primary objective was to assess the long-term safety of spesolimab in patients with hidradenitis suppurativa (HS), with additional objectives focusing on efficacy at a lower dose.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Period: Overall Study
Arm/Group | Prior Placebo (PP) | Prior Spesolimab (PS)
Started (Trial medication) | 15 | 30
Completed (Trial medication) | 7 | 9
Not Completed | 8 | 21
Not completed — Withdrawal by Subject | 1 | 10
Not completed — Lost to Follow-up | 2 | 4
Not completed — Lack of Efficacy | 0 | 2
Not completed — Adverse Event | 3 | 1
Not completed — Patient non-compliance | 0 | 1
Not completed — Personal reasons | 0 | 1
Not completed — Withdrawn as per protocol | 2 | 2

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set (SAF): The safety analysis set includes all participants who received at least one dose of the trial drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Prior Placebo (PP) | Prior Spesolimab (PS) | Total
Number analyzed (Participants) | 15 | 30 | 45
Age, Continuous [Mean (Standard Deviation); unit: Years] | 35.7 (10.7) | 35.5 (10.8) | 35.6 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 19 | 27
  Male | 7 | 11 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 14 | 25 | 39
  Unknown or Not Reported | 0 | 4 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 4 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 2 | 2 | 4
  White | 11 | 19 | 30
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 4 | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: TEAEs were defined as all adverse events (AEs) occurring from the start of treatment in this extension trial to the end of its residual effect period. AEs that began during the on-treatment period of the parent Proof of Concept and Confirmatory (PoCC) trial (1368-0052) and were still ongoing in this extension trial will also be considered as treatment-emergent.
Time Frame: From drug administration until the end of maintenance treatment period (120 weeks). This period includes the Residual effect period (REP) (i.e., 16 weeks after the last study treatment).
Population: Safety Analysis Set (SAF): This participant set included all participants who were enrolled and received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- Prior Placebo (PP): Participants in the placebo arm of the 1368-0052 Proof of Concept Clinical (PoCC) trial received an initial 1200 mg intravenous (i.v.) loading dose of spesolimab plus subcutaneous (s.c.) placebo at Visit 1, followed by 600 mg subcutaneous (s.c.) doses of spesolimab every two weeks for the next 12 weeks. Further dosing was based on changes in HS-PGA grade assessment from baseline to week 12.
Arm/Group | Prior Placebo (PP) | Prior Spesolimab (PS)
Number analyzed (Participants) | 15 | 30
Participants | 15 | 28

2. Secondary Outcome: Percent Change in Total Abscess and Inflammatory Nodule (AN) Count From Baseline up to Week 12
Description: Percentage change from baseline in total abscess and inflammatory nodule count at Week 12= [(Total Abscess at Week 12 + Total Inflammatory Nodule at Week 12) - (Total Abscess at baseline + Total Inflammatory Nodule at baseline)] *100/ (Total Abscess at baseline + Total Inflammatory Nodule at baseline).
  Percentage change from baseline in total abscess and inflammatory nodule count at Week 12 was modelled using a restricted maximum likelihood (REML)-based mixed effect model with repeated measures (MMRM) approach, accounting for the following sources of variation: fixed, categorical effects of treatment at each visit, prior use of TNF inhibitor and the fixed continuous effects of baseline at each visit (Weeks 1, 2, 4, 6, 8, 10, and 12) as well as random effect of each visit. Baseline refers to the last measurement prior to the start of spesolimab. The Least Squares Mean (Standard Error) of percentage change at Week 12 is reported.
Time Frame: MMRM included measurements from baseline (Week 12 of 1368-0052) and at Weeks 1, 2, 4, 6, 8, 10, and 12 after first drug administration.
Population: Safety Analysis Set (SAF): This participant set included all participants who received at least one dose of the study drug. Data up to the use of rescue therapy were included for analysis, and data post-use were censored. Only participants with non-missing endpoint data were included.
Measure: Least Squares Mean (Standard Error); unit: Percentage change
Arm/Group | Prior Placebo (PP) | Prior Spesolimab (PS)
Number analyzed (Participants) | 12 | 26
Percentage change | -18.3 (19.2) | -35.0 (12.7)

3. Secondary Outcome: Percentage Change in Total Draining Fistula (DF) Count From Baseline up to Week 12
Description: Percentage change from baseline in draining fistula at Week 12 was calculated as: [(total draining fistula at Week 12) - (total draining fistula at baseline)] * 100 %/ (total draining fistula at baseline). Percentage change from baseline in in draining fistula count at Week 12 was modelled using a restricted maximum likelihood (REML)-based mixed effect model with repeated measures (MMRM) approach, accounting for the following sources of variation: fixed, categorical effects of treatment at each visit, prior use of TNF inhibitor and the fixed continuous effects of baseline at each visit (Weeks 1, 2, 4, 6, 8, 10, and 12) as well as random effect of each visit.
  Baseline refers to the last measurement prior to the start of spesolimab. Unstructured covariance matrix was used.
Time Frame: MMRM included measurements from baseline (Week 12 of 1368-0052) and at Weeks 1, 2, 4, 6, 8, 10, and 12 after first drug administration. MMRM estimates of percentage change in draining fistula from baseline to Week 12 is reported.
Population: Safety Analysis Set (SAF): This patient set included all patients who received at least one dose of study drug. Data up to use of rescue therapy were included for analysis, and data post the use were censored. Only patients with baseline draining fistulas >=1 and non-missing endpoint data were included.
Measure: Least Squares Mean (Standard Error); unit: Percentage change
Arm/Group | Prior Placebo (PP) | Prior Spesolimab (PS)
Number analyzed (Participants) | 11 | 21
Percentage change | 25.4 (25.5) | -44.6 (18.1)

4. Secondary Outcome: Achievement of Hidradenitis Suppurativa Clinical Response (HiSCR) up to Week 12
Description: HiSCR is defined as at least a 50% reduction in the total abscess and inflammatory nodule (AN) count with no increase in abscess count and no increase in draining fistula count relative to baseline.
  Percentage of participants with achievement of Hidradenitis Suppurativa Clinical Response (HiSCR) at Week 12 is reported. Percentage of participants with achievement of HiSCR at Week 12 was calculated as: number of participants with achievement of HiSCR at Week 12/number of participants analyzed * 100.
Time Frame: At baseline (Week 0) and at Week 12.
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Prior Placebo (PP) | Prior Spesolimab (PS)
Number analyzed (Participants) | 12 | 27
Percentage of participants | 33.3 [13.8 to 60.9] | 40.7 [24.5 to 59.3]

5. Secondary Outcome: Change From Baseline in International Hidradenitis Suppurativa Severity Score System (IHS4) Value up to Week 12
Description: The IHS4 assesses the hidradenitis suppurativa (HS) severity and the resulting IHS4 score is arrived at by= number of nodules * 1 + number of abscesses * 2 + number of draining tunnels (fistulae or sinuses) * 4.
  A total score of 3 or less signifies mild, 4-10 signifies moderate and 11 or higher signifies severe disease.
  The minimum score is 0 while the maximum score is variable and depends on the counts of nodules, abscesses, and draining tunnels (fistulae or sinuses).
  Absolute change from baseline in IHS4 value at Week 12 was modelled using a restricted maximum likelihood (REML)-based mixed effect model with repeated measures (MMRM) approach, accounting for the following sources of variation: fixed, categorical effects of treatment at each visit, prior use of TNF inhibitor and the fixed continuous effects of baseline at each visit (Weeks 1, 2, 4, 6, 8, 10, and 12) as well as random effect of each visit. Baseline refers to the last measurement prior to the start of spesolimab.
Time Frame: MMRM included measurements at baseline (Week 0) and at Weeks 1, 2, 4, 6, 8, 10, and 12 after first drug administration. MMRM estimates of absolute change in IHS4 from baseline to Week 12 is reported.
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Prior Placebo (PP) | Prior Spesolimab (PS)
Number analyzed (Participants) | 13 | 26
Score on a scale | -3.1 (4.8) | -10.5 (3.3)

6. Secondary Outcome: Percentage of Participants With Hidradenitis Suppurativa Physician Global Assessment (HS-PGA) Score of 0 or 1 up to Week 12
Description: HS-PGA documents the physician's assessment of the participant's HS at a given timepoint. The HS-PGA score ranges from 0 to 5: 0=clear (no abscesses, draining fistula, inflammatory or noninflammatory nodules); 1=minimal (no abscesses, draining fistula, inflammatory nodules; noninflammatory nodules present); 2=mild (no abscesses, draining fistula, 1-4 inflammatory nodules; or 1 abscess or draining tunnel, no inflammatory nodules); 3=moderate (no abscesses, draining fistula, ≥5 inflammatory nodules; or 1 abscess/draining fistula, ≥1 inflammatory nodule; or 2-5 abscesses/draining fistula, <10 inflammatory nodules); 4=severe (2-5 abscesses/draining fistula, ≥10 inflammatory nodules); 5=very severe (>5 abscesses/draining fistula).
  The percentage of participants with HS-PGA 0 or 1 at Week 12 was calculated as: (number with HS-PGA 0/1 at Week 12 ÷ number analyzed) × 100.
Time Frame: At Week 12.
Population: Safety Analysis Set (SAF): This participant set included all participants who received at least one dose of study drug. Any binary data collected after use of any rescue therapy was censored and then imputed using the no response imputation (NRI) method as described in the statistical analysis plan.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Prior Placebo (PP) | Prior Spesolimab (PS)
Number analyzed (Participants) | 13 | 27
Percentage of participants | 0 [0 to 22.8] | 3.7 [0.7 to 18.3]

7. Secondary Outcome: Absolute Change From Baseline in Hidradenitis Suppurativa Area and Severity Index (HASI) Score up to Week 12
Description: The HASI assesses HS severity across four domains: erythema, induration, open ulcer, and draining fistula, scored on a 0 (none) to 3 (severe/extensive) Likert scale for each body region.
  For body surface area (BSA) assessment, the number of palms (one palm indicates 1% of the participant's BSA) involved for each body region (head, right axilla, left axilla, anterior chest, back, anterior bathing trunk, posterior bathing trunk, other) is assessed and converted to a percentage of that region. An area score was assigned to each region using the approach (0 = none, 1 = 1-9%, 2 = 10-29%, 3 = 30-49%, 4 = 50-69%, 5 = 70-89%, 6 = 90- 100%). Scores for the four domains of HS are summed and adjusted for the area affected, and the score of each area are summed to calculate the total HASI score, which ranges from 0 (no disease) to 72 (severe disease).
  The Least Squares Mean (Standard Error (SE)) was derived from mixed effect model with repeated measures (MMRM).
Time Frame: MMRM included measurements at baseline (Week 0) and at Weeks 1, 2, 4, 6, 8, 10, and 12 after first drug administration. MMRM estimates of absolute change from baseline in HASI score at Week 12 is reported.
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Prior Placebo (PP) | Prior Spesolimab (PS)
Number analyzed (Participants) | 13 | 26
Score on a scale | 5.0 (8.9) | -22.8 (6.1)

8. Secondary Outcome: Patients With Occurrence of at Least One Flare (Defined as at Least 25 % Increase in AN Count With a Minimum Increase of 2 Relative to Baseline) up to Week 12
Description: Percentage of participants with occurrence of at least one flare at Week 12. Flare was defined as at least 25 % increase in abscess and inflammatory nodule count with a minimum increase of 2 relative to baseline.
  Percentage of participants with occurrence of at least one flare at Week 12 was calculated as: number of participants with occurrence of at least one flare at Week 12/number of participants analyzed * 100.
Time Frame: Samples were taken at baseline (Week 0) and at Weeks 2, 4, 6, 8, 10, and 12 after first drug administration.
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Prior Placebo (PP) | Prior Spesolimab (PS)
Number analyzed (Participants) | 12 | 27
Percentage of participants | 8.3 [1.5 to 35.4] | 14.8 [5.9 to 32.5]

9. Secondary Outcome: Achievement of at Least 30% Reduction From Baseline in Numerical Rating Scale (NRS30) in Patient's Global Assessment of HS Pain up to Week 12
Description: The analysis assessed the percentage of participants who achieved at least a 30% reduction from baseline in the Numerical Rating Scale (NRS30) for the Participant's Global Assessment of HS Pain by Week 12.
  The HS Pain Numerical Rating Scale (NRS) measures HS-related pain severity, with a recall period of 24 hours and responses on an 11-point scale from 0 (no pain) to 10 (worst possible pain). For pain analysis, a weekly average of daily assessments was calculated at each visit, based on recorded values before the visit. Weeks with at least four reported daily values were included, ignoring any missing daily values.
  The percentage of participants achieving at least a 30% reduction from baseline in NRS30 by Week 12 was calculated as the number of participants meeting this criterion divided by the total number of participants analyzed * 100.
Time Frame: At baseline (Week 0) and at Week 12.
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Prior Placebo (PP) | Prior Spesolimab (PS)
Number analyzed (Participants) | 12 | 27
Percentage of participants | 25.0 [8.9 to 53.2] | 33.3 [20.2 to 55.5]

ADVERSE EVENTS:
Time Frame: All-cause mortality, AEs and SAEs: From drug administration until the end of maintenance treatment period (120 weeks). This period includes the Residual effect period (REP) (i.e., 16 weeks after the last study treatment).
Description: Safety Analysis Set (SAF): The safety analysis set includes all participants who received at least one dose of the trial drug.
Arm/Group | Prior Placebo (PP) | Prior Spesolimab (PS)
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/30
Serious Adverse Events (participants affected / at risk) | 4/15 | 6/30
Other Adverse Events (participants affected / at risk) | 15/15 | 27/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Prior Placebo (PP) (N=15) | Prior Spesolimab (PS) (N=30)
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Abdominal abscess (Infections and infestations) | 0 | 1
Acute hepatitis C (Infections and infestations) | 1 | 0
Latent tuberculosis (Infections and infestations) | 1 | 0
Vulval abscess (Infections and infestations) | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1
Guillain-Barre syndrome (Nervous system disorders) | 0 | 1
Acute psychosis (Psychiatric disorders) | 0 | 1
Hidradenitis (Skin and subcutaneous tissue disorders) | 1 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Prior Placebo (PP) (N=15) | Prior Spesolimab (PS) (N=30)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0
Ventricular extrasystoles (Cardiac disorders) | 1 | 0
Vision blurred (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 1 | 4
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Toothache (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 1 | 2
Axillary pain (General disorders) | 1 | 0
Chest pain (General disorders) | 1 | 1
Fatigue (General disorders) | 0 | 2
Feeling hot (General disorders) | 1 | 0
Influenza like illness (General disorders) | 0 | 3
Injection site bruising (General disorders) | 1 | 0
Injection site erythema (General disorders) | 1 | 2
Injection site haematoma (General disorders) | 1 | 2
Injection site pain (General disorders) | 0 | 2
Injection site pruritus (General disorders) | 0 | 2
Injection site swelling (General disorders) | 0 | 2
Pyrexia (General disorders) | 0 | 4
Swelling face (General disorders) | 1 | 0
Abscess sweat gland (Infections and infestations) | 1 | 0
Anal abscess (Infections and infestations) | 1 | 0
COVID-19 (Infections and infestations) | 1 | 13
Erythrasma (Infections and infestations) | 1 | 1
Gastroenteritis (Infections and infestations) | 0 | 3
Gastroenteritis viral (Infections and infestations) | 1 | 1
Influenza (Infections and infestations) | 1 | 1
Nail infection (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 3 | 4
Pilonidal disease (Infections and infestations) | 0 | 2
Sinusitis (Infections and infestations) | 0 | 2
Subcutaneous abscess (Infections and infestations) | 1 | 0
Tinea cruris (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 2
Vulvovaginal mycotic infection (Infections and infestations) | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 1
Sunburn (Injury, poisoning and procedural complications) | 1 | 0
Amylase increased (Investigations) | 1 | 0
Bacterial test positive (Investigations) | 1 | 0
Blood fibrinogen increased (Investigations) | 1 | 1
Blood pressure increased (Investigations) | 1 | 0
C-reactive protein increased (Investigations) | 1 | 1
Haemoglobin decreased (Investigations) | 1 | 0
Heart rate irregular (Investigations) | 1 | 0
Hepatic enzyme increased (Investigations) | 1 | 1
Lipase increased (Investigations) | 1 | 0
Mycobacterium test positive (Investigations) | 1 | 0
Platelet count increased (Investigations) | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 2
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 3
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 6
Fistula (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 4
Sacral pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 2
Headache (Nervous system disorders) | 1 | 4
Lethargy (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 2
Anxiety (Psychiatric disorders) | 1 | 0
Leukocyturia (Renal and urinary disorders) | 1 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 1 | 2
Heavy menstrual bleeding (Reproductive system and breast disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Acne (Skin and subcutaneous tissue disorders) | 0 | 2
Eczema (Skin and subcutaneous tissue disorders) | 1 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Hidradenitis (Skin and subcutaneous tissue disorders) | 8 | 10
Intertrigo (Skin and subcutaneous tissue disorders) | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Rosacea (Skin and subcutaneous tissue disorders) | 1 | 1
Skin haemorrhage (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2022-07-04): https://cdn.clinicaltrials.gov/large-docs/91/NCT04876391/Prot_000.pdf
  • Statistical Analysis Plan (2024-06-04): https://cdn.clinicaltrials.gov/large-docs/91/NCT04876391/SAP_001.pdf